CLINICAL TRIAL: NCT00766792
Title: Removal of Uremic Toxins With Nocturnal Dialysis Versus Standard Dialysis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Raymond Vanholder, University Hospital Ghent
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2005/288
Record Dates: First submitted 2008-10-03; First posted 2008-10-06 (Estimated); Last update posted 2008-10-31 (Estimated); Status verified 2008-10

CONDITIONS: Chronic Renal Failure
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Nocturnal dialysis
  Interventions: Procedure: Nocturnal dialysis
- 2 (Active Comparator): Standard dialysis
  Interventions: Procedure: Standard dialysis

INTERVENTIONS:
Procedure: Nocturnal dialysis — Switch to nocturnal dialysis (3 times 480 min/week)
  Arms: 1
Procedure: Standard dialysis — Standard dialysis (3 times 240-270 min/week)
  Arms: 2

SUMMARY:
Dialysis patients, who decide to switch from standard dialysis (3 times 240-270 min/week) to nocturnal dialysis (3 times 480 min/week), will be followed. In parallel a control group with patients staying on standard dialysis will be followed. The study will last 30 weeks. During this period blood samples (pre- and post-dialysis: 10 times; inlet and outlet of dialyzer: 3 times) will be collected on predetermined time points. Concentration of several uremic retention solutes will be determined.

ELIGIBILITY:
Inclusion Criteria:

* age > 18 years

Exclusion Criteria:

* pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2005-12; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
To evaluate what is more effective for removal of uremic toxins - nocturnal versus standard dialysis? | 30 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Raymond Vanholder, MD, PhD, Principal Investigator — University Hospital, Ghent
Locations (1):
- University Hospital Ghent, Ghent, Belgium

REFERENCES:
- See also: Website of the University Hospital Ghent — http://www.uzgent.be